CLINICAL TRIAL: NCT00406679
Title: Single-Dose Comparison of the Analgesic Efficacy, Safety and Tolerability of Two Paracetamol 1%-Containing Solutions and Placebo in a Post-Surgical Dental Pain Model
Brief Title: Analgesic Efficacy, Safety and Tolerability of Two Paracetamol-containing Solutions in Post-Surgical Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Keyvan Tadjalli Mehr, MD, Baxter Healthcare Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-01270-A015; EudraCT2005-005575-14
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Pain, Postoperative
Keywords: pain, postoperative; surgery, oral; surgery, dental
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Paracetamol (acetaminophen) solution experimental
- 2 (Placebo Comparator)
  Interventions: Drug: placebo
- 3 (Active Comparator)
  Interventions: Drug: paracetamol (acetaminophen) solution commercial

INTERVENTIONS:
Drug: Paracetamol (acetaminophen) solution experimental — 1 gm IV
  Other Names: paracetamol; acetaminophen
  Arms: 1
Drug: paracetamol (acetaminophen) solution commercial — 1 gm IV
  Other Names: paracetamol; acetaminophen
  Arms: 3
Drug: placebo — equivalent volume IV 0.9% sodium chloride (equivalent volume)
  Other Names: sodium chloride; saline
  Arms: 2

SUMMARY:
The aim of the study is to evaluate the therapeutic efficacy and safety of two different paracetamol-containing solutions in postoperative dental pain. They will be compared to placebo (a dummy treatment which contains no active ingredient).

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II and scheduled for elective surgical extraction of 1 or more impacted mandibular 3rd molars, at least 1 of which must be a fully or partially impacted mandibular 3rd molar requiring mandibular bone removal.
* Moderate or severe pain within 4 hours after the completion of surgery.

Exclusion Criteria:

* Another acute or chronic painful physical condition
* Use of any other analgesics (within 24 hours), sedatives, or narcotic drugs as well as microsomal enzyme inducers
* Inability to use and understand Visual Analog Scale and Verbal Rating Score

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Tadjalli-Mehr, MD, Study Director — Baxter Healthcare Corporation
Locations (2):
- United Kingdom (2):
  - University Dental Hospital of Manchester, Manchester, England
  - University Dental Hospital NHS Trust Cardiff, Cardiff, Wales